CLINICAL TRIAL: NCT06803849
Title: Association of Heterogeneous Circulating Biomarkers and Anamnestic Factors of Pregnancy Adverse Course and Outcomes With the Prognosis of Heart Failure With Preserved Ejection Fraction
Acronym: CARPO-HF
Status: Recruiting | Type: Observational
Sponsor: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Responsible Party: Sponsor
Other Study IDs: 04-07/24
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure With Preserved Ejection Fraction (HFPEF)
Keywords: Heart Failure with Preserved Ejection Fraction; Adverse Pregnancy Outcomes; Gestational Hypertension; Preeclampsia; Gestational Diabetes Mellitus; Heart Diseases; Cardiovascular Diseases; Heart Failure; Pregnancy Complications; Preterm delivery; Stillbirth
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia; Diabetes, Gestational; Heart Diseases; Cardiovascular Diseases; Heart Failure; Pregnancy Complications; Premature Birth; Stillbirth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with anamnestic factors of pregnancy adverse course and outcomes
- Patients without anamnestic factors of pregnancy adverse course and outcomes

SUMMARY:
The primary purpose of this study is to evaluate possible association of some heterogeneous circulating biomarkers and anamnestic factors of pregnancy adverse course and outcomes with the prognosis of heart failure with preserved ejection fraction. The study population includes women aged 60-74 years with history of pregnancy with duration at least 20 weeks and diagnosed heart failure with preserved ejection fraction based on algorithm HFA-PEFF.

The following pregnancy complications are assessed on the initial visit: gestational hypertension, preeclampsia, gestation diabetes mellitus and recently introduced as cardiovascular disease risk factors preterm delivery, stillbirth, miscarriage. This information is collected through a questionnaire which additionally includes questions about menopause and the circumstances of its onset. The data about comorbidities, results of laboratory and instrumental tests is collected from medical records. After the interview short physical examination is performed to measure anthropometric data and objective signs of congestion. In addition, medical Research Council Scale survey is conducted to assess the subjective severity of shortness of breath and a six-minute walking test to objectively evaluate the heart failure functional class.

After inclusion in the study blood sampling is performed to measure the concentration of a number of biomarkers which are recognized as prognostically significant in context of heart failure: high-sensitivity troponin I, soluble suppression of tumorigenicity 2 protein, heat shock protein 27, cystatin C. As part of the study echocardiography is also performed with evaluation of left ventricular global longitudinal strain and left atrial strain to assess systolic and diastolic myocardium function.

12 months after the initial visit, participants are contacted by telephone. The data about newly diagnosed chronic non-communicable diseases, emergency hospitalization for any cause and major adverse cardiovascular events is collected. If there is no response from the research participant, the cause, including possible hospitalization or death, is determined by telephone contact with the participant's trusted person.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 60-74 years
* Heart failure with preserved ejection fraction (diagnosed by using HFA-PEFF algorithm)
* History of pregnancy with duration at least 20 weeks
* Willing and legally able to sign informed consent

Exclusion Criteria:

* History of ejection fraction less than 50% diagnosed by echocardiography
* Diagnosed cognitive impairment or dementia
* The state of cardiovascular disease decompensation
* Exacerbation of comorbidities
* The presence of chronic diseases that may affect the results of the study: ischemic heart disease (unstable angina, stable effort angina III-IV grade, previous myocardial infarction), previous Ischemic/hemorrhagic stroke, severe valvular heart diseases, cardiomyopathy, myocarditis, uncontrolled bronchial asthma or chronic obstructive pulmonary disease, terminal chronic kidney disease requiring dialysis, implanted pacemaker (including cardiac resynchronisation device, or defibrillator), active cancer, history of chemotherapy or radiation therapy to the chest area

Ages: 60 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged 60-74 years with history of pregnancy with duration at least 20 weeks and diagnosed heart failure with preserved ejection fraction based on algorithm HFA-PEFF
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Combined endpoint made up of emergency hospitalization for any cause, major adverse cardiovascular events and all-cause mortality | From the date of enrollment until the date of the first emergency hospitalization for any cause or date of any major adverse cardiovascular event or all-cause death, whichever came first, assessed up to 1 years
  Major adverse cardiovascular events include myocardial infarction, stroke, cardiovascular death

SECONDARY OUTCOMES:
Newly diagnosed chronic non-communicable disease | From the date of enrollment until the date of diagnosis of any chronic non-communicable disease, whichever came first, assessed up to 1 years
  Chronic non-communicable diseases include cardiovascular diseases, respiratory system diseases, diabetes mellitus, cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Federal State Budgetary Institution National Medical Research Center for Therapy and Preventive Medicine of the Ministry of Healthсare of the Russian Federation, Moscow, Russia